CLINICAL TRIAL: NCT04080375
Title: the Effectiveness of Preoperative Vaginal Dinoprostone in Reducing Blood Loss During Abdominal Myomectomy:a Randomized Controlled Trial
Brief Title: Preoperative Vaginal Dinoprostone Prior to Abdominal Myomectomy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Samy aly ashour, assistant professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: dinoprostone myomectomy
Record Dates: First submitted 2019-09-04; First posted 2019-09-06 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Myomectomy
MeSH Terms: interventions — Dinoprostone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dinoprostone 3 mg (Experimental): patients will take 1 tablet of vaginal dinoprostone 1 hour before the surgery
  Interventions: Drug: Dinoprostone 3 mg
- placebo (Placebo Comparator): patients will take 1 tablet of placebo 1 hour before the surgery
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Dinoprostone 3 mg — the patient will take one vaginal tablet of 3 mg dinoprostone 1 hour before surgery
  Arms: dinoprostone 3 mg
Drug: placebo — the patient will take one vaginal tablet of placebo 1 hour before surgery
  Arms: placebo

SUMMARY:
The aim of the study is to compare the effectiveness of vaginal dinoprostone 3 mg versus placebo before myomectomy to decrease blood loss during and after the operation.

ELIGIBILITY:
Inclusion Criteria:

* • Patients presenting for abdominal myomectomy with documented uterine fibroids on pelvic imaging

  * Age ≥ 18 years and ≤ 50 years
  * Pre-operative hemoglobin >8 g/dl
  * Ability to understand and the willingness to sign a written informed consent.
  * Admissible medical/surgical history
  * Five or less symptomatic uterine myomas
  * All myomas are subserous or intramural.
  * Uterine size less than 24 weeks pregnancy

Exclusion Criteria:

* • Patients who have had a prior abdominal myomectomy

  * Post-menopausal women
  * Patients with known bleeding/clotting disorders
  * Patients with a history of gynecologic malignancy
  * Hypertension.
  * Cardiac and Pulmonary diseases.
  * Obesity (body mass index > 30 kg/m2).
  * History of allergic reactions attributed to misoprostol
  * Cases that will require intraoperative conversion of myomectomy to hysterectomy.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 100 (Estimated)
Dates: Start 2019-09-10 (Estimated); Primary Completion 2019-11-30 (Estimated); Study Completion 2019-12-10 (Estimated)

PRIMARY OUTCOMES:
Mean amount of intraoperative blood loss | intraoperative
  Mean amount of intraoperative blood loss in ml

SECONDARY OUTCOMES:
Change of hemoglobin after surgery | 24 hours
  Change of hemoglobin(g/dl) after surgery

CONTACTS AND LOCATIONS:
Overall Officials: AHMED SAMY, Principal Investigator — Cairo University